CLINICAL TRIAL: NCT00713583
Title: Contingency Management Plus Levodopa/Carbidopa for Treatment of Cocaine Dependence
Brief Title: Carbidopa/Levodopa Combined With Behavioral Therapy for the Treatment of Cocaine Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Joy Schmitz, Professor - Psychiatry, Behavioral Sciences, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R01DA023608-01 (NIH); 1R01DA023608-01 (NIH); R01DA023608-01 (NIH); DPMCDA (Other: NIDA)
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Results first posted 2018-03-19 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-03

CONDITIONS: Cocaine Dependence
Keywords: Cocaine, levodopa, contingency management
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Levodopa; carbidopa, levodopa drug combination; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Levodopa pharmacotherapy (Experimental): Levodopa pharmacotherapy (800mg levodopa and 200mg carbidopa per day), cognitive behavioral therapy (CBT), and contingency management (CM).
  Interventions: Drug: levodopa; Behavioral: Cognitive Behavioral Therapy; Behavioral: Contingency Management
- Placebo (Placebo Comparator): Placebo, cognitive behavioral therapy (CBT), and contingency management (CM).
  Interventions: Drug: Placebo; Behavioral: Cognitive Behavioral Therapy; Behavioral: Contingency Management

INTERVENTIONS:
Drug: levodopa — 800mg levodopa and 200mg carbidopa per day
  Other Names: Sinemet
  Arms: Levodopa pharmacotherapy
Drug: Placebo — Placebo
  Arms: Placebo
Behavioral: Cognitive Behavioral Therapy — Participants received individual cognitive behavioral therapy (CBT) in 50-minute weekly sessions. These sessions were manual-driven and based on the relapse prevention model proposed by Marlatt and Gordon (1985). Trained masters-level therapists, under the supervision of senior therapists and the principal investigator, worked with participants to teach them how to recognize and cope with risky situations that could influence their cocaine use through self-monitoring of situational craving and drug use stimuli, coping skills training, and lifestyle modifications.
Behavioral: Contingency Management — An abstinence-based contingency management (CM) procedure was used. Participants earned vouchers according to the reward schedule recommended by Budney and Higgins (1998), beginning at $2.50 for the first cocaine-negative urine. For each consecutive cocaine-negative urine, voucher values increased by $1.25 with a $10 bonus given for provision of three consecutive cocaine-negative urines within a week. A cocaine-positive urine or failure to provide a scheduled urine sample resulted in a reset of the schedule to the initial value of $2.50. After provision of five negative urines, the voucher returned to the value prior to the reset. Participants were able to redeem their vouchers for small amounts of cash (≤$25) or gift cards for goods and services.

SUMMARY:
Cocaine dependence is a major public health problem and the development of a treatment for this disorder is a priority. To date, treatment interventions based on positive incentive principles have shown the strongest effects for improving substance use outcomes. One such example is contingency management (CM) interventions in which nondrug rewards are used to compete with cocaine. Recent evidence suggests that certain medications improve response to CM interventions, particularly agents that target dopamine reward systems in the brain. A promising dopamine-enhancing medication is levodopa. The study team has observed the strongest effects of levodopa when the medication is administered in the context of CM therapy, perhaps through mechanisms that enhance reward saliency. The proposed study is designed to further evaluate this promising treatment approach. Cocaine dependent outpatients will participate in a randomized, 2-group (levodopa vs. placebo), double-blind clinical trial. CM will be behavioral therapy platform for both treatment groups. The study will test the primary hypothesis that CM+levodopa will be more effective than CM+placebo in reducing cocaine use. This study is expected to validate the usefulness of a new behavioral-pharmacological treatment approach for cocaine dependence.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 60 years of age
* meet Diagnostic and Statistical Manual of Mental Disorders, 4th. Edition (DSM-IV) criteria for current cocaine dependence.
* be in acceptable health on the basis of interview, medical history and physical exam.

Exclusion Criteria:

* current DSM-IV diagnosis of any psychoactive substance dependence other than cocaine, marijuana, or nicotine.
* have a DSM-IV axis I psychiatric disorder or neurological disease or disorder requiring ongoing treatment and/or making study participation unsafe.
* have significant current suicidal or homicidal ideation.
* have medical conditions contraindicating levodopa/carbidopa pharmacotherapy. Conditions include severe pulmonary disease (bronchial asthma, emphysema), cardiovascular disease (severe or history of myocardial infarction with residual arrhythmias), narrow angle glaucoma, melanoma, history of peptic ulcer, renal function impairment.
* taking medications known to have significant drug interactions with levodopa/carbidopa (e.g., monoamine oxidase (MAO) inhibitors, anticonvulsants, haloperidol, phenothiazines, selegiline, anesthetics).
* currently or recently (last 3 months) treated for substance use or another psychiatric condition.
* having conditions of probation or parole requiring reports of drug use to officers of the court.
* impending incarceration.
* pregnant or nursing for female patients.
* inability to read, write, or speak English.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2008-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joy M Schmitz, PhD, Principal Investigator — University of Texas at Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Levodopa Pharmacotherapy: Levodopa pharmacotherapy, cognitive behavioral therapy (CBT), and contingency management (CM).
Period: Overall Study
Arm/Group | Levodopa Pharmacotherapy | Placebo
Started | 45 | 40
Completed | 45 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levodopa Pharmacotherapy | Placebo | Total
Number analyzed (Participants) | 45 | 40 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (7.9) | 45 (9.2) | 46 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 15
  Male | 35 | 35 | 70
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45 | 40 | 85

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Abstinence From Cocaine as Assessed by Treatment Effectiveness Score (TES)
Description: The Treatment Effectiveness Score (TES) is the number of cocaine-negative urines collected out of the total scheduled urine tests for the 12-week trial (36 total scheduled urine tests per participant). The mean number of cocaine-negative urines over all time points is reported in this outcome measure.
Time Frame: 12 weeks of treatment
Measure: Mean (Standard Deviation); unit: cocaine-negative urines
Arm/Group | Levodopa Pharmacotherapy | Placebo
Number analyzed (Participants) | 45 | 40
cocaine-negative urines | 7 (11.7) | 9 (12.6)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Levodopa Pharmacotherapy | Placebo
Serious Adverse Events (participants affected / at risk) | 6/45 | 3/40
Other Adverse Events (participants affected / at risk) | 0/45 | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levodopa Pharmacotherapy (N=45) | Placebo (N=40)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Photosensitivity (Eye disorders) | 1 (1) | 0 (0)
Head injury (General disorders) | 1 (1) | 0 (0)
Suicide ideation (Psychiatric disorders) | 0 (0) | 1 (1)
abscess (Infections and infestations) | 0 (0) | 1 (1)
Transient inability to speak (General disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Vascular disorders) | 0 (0) | 1 (1)
Blood clot (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Lower than expected rates of retention and medication compliance likely reduced the statistical power of the study for estimating treatment effects of the medication intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes